CLINICAL TRIAL: NCT00163397
Title: A Comparative Study of Inhaled Ciclesonide 160 mcg/Day vs Budesonide 400 mcg/Day in Patients With Asthma
Brief Title: Efficacy of Ciclesonide Versus Budesonide in Patients With Asthma (18 to 75 y) (BY9010/M1-137)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BY9010/M1-137
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-10

CONDITIONS: Asthma
Keywords: Asthma; Ciclesonide; Budesonide
MeSH Terms: conditions — Asthma | interventions — ciclesonide

INTERVENTIONS:
Drug: Ciclesonide

SUMMARY:
The aim of the study is to investigate the efficacy of ciclesonide versus budesonide on lung function, symptoms and use of rescue medication in patients with asthma. Ciclesonide and budesonide will be inhaled once daily at one dose level each. The study duration consists of a baseline period (1 to 4 weeks) and a treatment period (12 weeks). The study will provide further data on safety and tolerability of ciclesonide.

ELIGIBILITY:
Main Inclusion Criteria:

* During the last 4 weeks prior to baseline, treatment with an inhaled steroid (dosage: up to 250 mcg fluticasone propionate or equivalent)
* FEV1 80 - 105% of predicted
* Healthy with the exception of asthma
* Written informed consent has been obtained
* Outpatients
* Patients who have a history of persistent bronchial asthma for at least 6 months

Main Exclusion Criteria:

* Concomitant severe diseases or diseases which are contraindications for the use of inhaled steroids
* Concomitant COPD (i.e. chronic bronchitis or emphysema) and/or other relevant lung diseases causing alternating impairment in lung function
* An asthma exacerbation or an infection of the lower airways prior to entry into the baseline period
* Pregnancy
* Intention to become pregnant during the course of the study
* Breast feeding
* Lack of safe contraception
* Patient is current smoker with 10 or more pack-years
* Patient is ex-smoker with 10 or more pack-years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2004-01; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
FEV1 absolute values.

SECONDARY OUTCOMES:
FEV1 as percent of predicted
FVC
PEF absolute values
morning and evening PEF from diary
diurnal PEF fluctuation
asthma symptom score from diary
use of rescue medication from diary
number of symptom free- and rescue medication free days
dropout rate due to asthma exacerbations
time until first asthma exacerbation
number of days with asthma control
onset of effect
subgroup analysis for ex/current smokers and non-smokers
AQLQ(S)
physical examination
vital signs
laboratory work-up
adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca AstraZeneca, Study Director — AstraZeneca
Locations (3):
- Malaysia (2):
  - Altana Pharma/Nycomed, Kota Bharu / Kelantan
  - Altana Pharma/Nycomed, Kuala Lumpur
- Altana Pharma/Nycomed, Taipei, Taiwan

REFERENCES:
- See also: BY9010-M1-137-RDS-2006-12-03.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=4522&filename=BY9010-M1-137-RDS-2006-12-03.pdf